CLINICAL TRIAL: NCT05818761
Title: The Effects of Virtual Reality and Stress Ball Distraction on Procedure-Related Emotional Appearance, Pain, Fear, and Anxiety During Phlebotomy in Children
Brief Title: Distraction on Procedure-Related Emotional Appearance, Pain, Fear, and Anxiety During Phlebotomy in Children
Acronym: VR-DEU22
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Gülçin Özalp Gerçeker, pHD, Assoc. Prof., Dokuz Eylul University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: VR-DEU22
Record Dates: First submitted 2023-03-30; First posted 2023-04-19 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Pain, Acute; Fear; Anxiety State
MeSH Terms: conditions — Acute Pain; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomised
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- virtual reality (Experimental): watching the application by wearing virtual glasses to the child during the phlebotomy
  Interventions: Device: virtual reality
- Stress ball (Experimental): a stress ball will be given to the child's hand, and he will be asked to squeeze continuously before the blood draw attempt begins, and to continue squeezing during the procedure.
  Interventions: Behavioral: stress ball
- control (No Intervention): standard approach

INTERVENTIONS:
Device: virtual reality — wearing virtual reality glasses
  Arms: virtual reality
Behavioral: stress ball — squeezing the stress ball during the attempt
  Arms: Stress ball

SUMMARY:
This randomized controlled study was planned to evaluate the effects of distraction methods, using virtual reality or a stress ball, on the emotional appearance, pain, fear, and anxiety associated with the procedure, during the phlebotomy in children aged 6-12 in a private blood collection unit.

DETAILED DESCRIPTION:
H1: There is a difference between the groups in terms of pain, fear, anxiety and emotional appearance scores related to the intervention during the blood draw attempt.

A standard approach will be applied to all children. Standard approach; giving information about the procedure, the nurse introducing herself, choosing the area together, being with the parent and talking to the child during the procedure, "I'm starting now, I'm cleaning the area, take a deep breath, I'm applying it now, it may hurt a little, you shouldn't move, it will take a very short time, I will cover it with tape " contains.

In the virtual reality glasses group, a tourniquet will be attached to the extremity where the intervention will be performed. By wearing virtual glasses, the video will be started.

In the stress ball group, before the intervention is applied, the other hand will be given a stress ball and asked to squeeze it.

In the control group, communication with the child will continue during the intervention with the questions mentioned above.

When the nurse decides on the area where the PICT will be performed (the minute will be recorded), she will use the words "I am cleaning the area, take a deep breath, now I am applying the injection, it may hurt a little, you should not move, it will be very short".

The intervention will be stopped when the blood draw attempt fails in all groups.

5 minutes after the blood draw attempt, the child will be asked to rate the most painful moment felt during the procedure using the Facial Expressions Rating Scale. The Child Fear Scale (CDS) and Child Anxiety Scale-State (CAS-D) will be given to the child to assess how anxious and frightened he is during the procedure. The child will be asked to mark with a pencil. The Emotional Appearance Scale for Children will be evaluated by the nurse after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* The age range of children is between 6-12
* The child's consent to voluntarily participate in the study
* Parent's willingness to participate in the study voluntarily
* Obtaining consent forms from child and parent

Exclusion Criteria:

* The child has a physical or psychological deficit that would prevent them from wearing glasses to watch virtual reality.
* fever (>37.5C) and severe dehydration
* The child takes analgesics before the blood draw
* Wearing glasses

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 150 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-10 (Actual)

PRIMARY OUTCOMES:
Pain assesed by Wong-Baker FACES | up to 5 minutes after the phelobotomy
  Wong-Baker FACES (WB-FACES) Pain Rating Scale used. This scale uses in children aged 3 and older to rate pain severity. This numeric rating scale ranges from 0 to 10. Faces show emotions from smiling (0 = very happy/ no pain) to crying (10 = hurts worst).
Anxiety assesed by Children Anxiety Meter-State | up to 5 minutes after the phelobotomy
  The Children's Anxiety Meter (CAM-S). The Children's Anxiety Meter assesses children's anxiety and uses before medical procedures. This scale is drawn like a thermometer with a bulb at the bottom and also includes horizontal lines at intervals going up to the top (0-10). This scale ranges from 0 to 10. Higher values represent higher anxiety
Fear assesed by Child Fear Scale | up to 5 minutes after the phelobotomy
  The Child Fear Scale (CFS). The Child Fear Scale will use.This one-item scale measures procedure-related fear in children, consists of five sex-neutral faces, ranges from 0 (no fear) to extreme fear. This rating scale ranges from 0 to 4. It ranges from a no fear (neutral) face (0) on the far left to a face showing extreme fear on the far right. Higher scores mean a worse outcome. The rater responds indicates the level of fear. It can be used during the procedure for children aged 5-10 years.

SECONDARY OUTCOMES:
Emotional Appearance | up to 5 minutes after the phelobotomy
  Emotional Appearance Scale for Children will use. This scale allows direct behavioral observation, consists of 5 different behavioral categories; 'Facial Expression', 'Speaking', 'Activity', 'Interaction' and 'Cooperation Level'. Scale scoring is done by reviewing the descriptions of behavior in each category and selecting the numerical value that most represents the observed behavior. Each category is scored from 1 to 5.

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin Özalp Gerçeker, pHD, Principal Investigator — Dokuz Eylul University
Locations (1):
- Gülçin Özalp Gerçeker, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gerceker GO, Bektas I, Yardimci F. The effects of virtual reality and stress ball distraction on procedure-related emotional appearance, pain, fear, and anxiety during phlebotomy in children: A randomized controlled study. J Pediatr Nurs. 2024 Nov-Dec;79:197-204. doi: 10.1016/j.pedn.2024.08.029. Epub 2024 Sep 17. PMID 39293201